CLINICAL TRIAL: NCT04030325
Title: Motivating Campus Change Study
Acronym: MC2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Mary Larimer, Professor, School of Medicine: Psychiatry And Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007499; R37AA012547-11A1 (NIH)
Record Dates: First submitted 2019-06-05; First posted 2019-07-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Drinking Behavior
MeSH Terms: conditions — Drinking Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Sequential Post Feedback Information Delivery (Experimental): Participants receive the first component of their PFI immediately following Baseline and subsequently receive 1 component each week until they receive all 4 components. Participants will complete a Post Feedback Survey and a 3 week follow back and Knowledge assessment.
  Interventions: Behavioral: Sequential Personalized Feedback Intervention Delivery
- Sequential Post Feedback Information Delivery +Text Messages (Experimental): Participants receive the first component of their PFI immediately following Baseline and subsequently receive 1 component each week until they receive all 4 components. Participants will complete a Post Feedback Survey and a 3 week follow back and Knowledge assessment. Additionally, participants receive the Text Message Booster Component in the days before and during the high risk drinking event celebration(s).
  Interventions: Behavioral: Sequential Personalized Feedback Intervention Delivery; Behavioral: Text Message Boosters
- Simultaneous Post Feedback Information Delivery (Experimental): Participants receive all 4 feedback components immediately after providing consent to the Pilot Feasibility Study following the Screening/Baseline Survey. Participants complete a brief 10 minute Post-Feedback Survey and a 3 Week Followup Survey to assess knowledge of the intervention feedback content.
  Interventions: Behavioral: Simultaneous Personalized Feedback Intervention Delivery
- Simultaneous Post Feedback Information Delivery +Text Messages (Experimental): Participants receive all 4 feedback components immediately after providing consent to the Pilot Feasibility Study following the Screening/Baseline Survey. Participants complete a brief 10 minute Post-Feedback Survey and a 3 Week Followup Survey to assess knowledge of the intervention feedback content. Additionally, participants receive the Text Message Booster Component in the days before and during the high risk drinking event celebration(s).
  Interventions: Behavioral: Simultaneous Personalized Feedback Intervention Delivery; Behavioral: Text Message Boosters
- Assessment Only Control (No Intervention): Participants complete baseline survey, longitudinal follow up assessments, and pre- and post- event surveys.

INTERVENTIONS:
Behavioral: Sequential Personalized Feedback Intervention Delivery — Sequential PFI delivery over 3 weeks after baseline survey
  Arms: Sequential Post Feedback Information Delivery; Sequential Post Feedback Information Delivery +Text Messages
Behavioral: Simultaneous Personalized Feedback Intervention Delivery — Simultaneous PFI delivery after baseline survey
  Arms: Simultaneous Post Feedback Information Delivery; Simultaneous Post Feedback Information Delivery +Text Messages
Behavioral: Text Message Boosters — Text message boosters on PFI content during week of high risk drinking events
  Arms: Sequential Post Feedback Information Delivery +Text Messages; Simultaneous Post Feedback Information Delivery +Text Messages

SUMMARY:
The study evaluates the relative merit of a multi-component PFI presented in the traditional simultaneous delivery (i.e., all components at once) versus a sequential format, wherein individual PFI components are delivered one at a time over several weeks to minimize time and attention demands for each component.

DETAILED DESCRIPTION:
This study builds upon the latest alcohol intervention literature to develop and test the next wave of personalized feedback interventions (PFIs) to address harmful alcohol use among college students. The purpose of this research is to determine optimal configuration of PFIs to take advantage of the clarity and initial impact of single-component PFIs and greater effect size and duration of personalized multi-component PFIs. The Investigators seek to increase and evaluate engagement with the PFI and text-message materials and boost innovation of both content and process of the intervention. In addition to PFI content and delivery, the investigators will use qualitative and quantitative methods to determine personal relevance of the chosen high-risk events among a sample of students who engage in heavy episodic drinking to better understand duration of PFI effects impacted by fluctuations in drinking associated with high-risk events. Prior interventions have targeted drinking in general or a single high-risk drinking event (e.g., Spring Break), but have not targeted both general and event-specific drinking together. These enhanced intervention effects, could have a significant impact on risks associated with college student drinking, and can be rapidly disseminated and implemented on campuses nationwide to address the public health problem posed by heavy episodic drinking among college students.

ELIGIBILITY:
Inclusion Criteria:

* at least 1 heavy episodic drinking episode in the past month
* at least 3 negative alcohol related consequences on Rutgers Alcohol Problem Index/ Young Adult Alcohol Problems Screening Test in the past 3 months for cohort 1
* at least 2 negative alcohol related consequences on Rutgers Alcohol Problem Index/ Young Adult Alcohol Problems Screening Test in the past month for cohort 2 - 5
* Indicate they own a cell phone with text message capabilities and consent to receiving text messages

Exclusion Criteria:

* Doesn't meet inclusion criteria
* Unwillingness to participate
* Failure to provide consent
* Plan to travel internationally in the next 12 months (for intervention text purposes)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1012 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Alcohol Use at 6 months | 6 months of assessment
  The first primary outcome of this program of research is to assess change in alcohol use from baseline to 6 months utilizing the Daily Drinking Questionnaire. The Daily Drinking Questionnaire assesses typical number of drinks on each of day of a typical week in the past month.
  Participants are allowed to enter the number of drinks for each day of the week. Values for each day will be summed together to create a composite score of typical weekly drinking. Minimum value is zero (0) and there is no maximum for the scale. Data will be assessed for outliers.
Change from Baseline Alcohol Use at 12 months | 12 months of assessment
  The second primary outcome of this program of research is to assess change in alcohol use from baseline to 12 months utilizing the Daily Drinking Questionnaire. The Daily Drinking Questionnaire assesses typical number of drinks on each of day of a typical week in the past month.
  Participants are allowed to enter the number of drinks for each day of the week. Values for each day will be summed together to create a composite score of typical weekly drinking. Minimum value is zero (0) and there is no maximum for the scale. Data will be assessed for outliers.
Change from Baseline Alcohol Use at 18 months | 18 months of assessment
  The third primary outcome of this program of research is to assess change in alcohol use from baseline to 18 months utilizing the Daily Drinking Questionnaire. The Daily Drinking Questionnaire assesses typical number of drinks on each of day of a typical week in the past month.
  Participants are allowed to enter the number of drinks for each day of the week. Values for each day will be summed together to create a composite score of typical weekly drinking. Minimum value is zero (0) and there is no maximum for the scale. Data will be assessed for outliers.
Change from Baseline Alcohol Use at 24 months | 24 months of assessment
  The fourth primary outcome of this program of research is to assess change in alcohol use from baseline to 24 months utilizing the Daily Drinking Questionnaire. The Daily Drinking Questionnaire assesses typical number of drinks on each of day of a typical week in the past month.
  Participants are allowed to enter the number of drinks for each day of the week. Values for each day will be summed together to create a composite score of typical weekly drinking. Minimum value is zero (0) and there is no maximum for the scale. Data will be assessed for outliers.

SECONDARY OUTCOMES:
Alcohol Use on New Years Eve | 2 days
  We will assess differences between arms on alcohol use on New Year's Eve and New Year's Day
Alcohol Use during Spring Break | 10 days
  We will assess differences between arms on alcohol use during the 10 days of Spring Break
Alcohol Use on 4th of July | 4 days
  We will assess differences between arms on alcohol use during 4 days surrounding 4th of July
Alcohol Use on Halloween | 4 days
  We will assess differences between arms on alcohol use during 4 days surrounding Halloween
Alcohol Use during Birthday | 10 days
  We will assess differences between arms on alcohol use during 10 days surrounding the participant's birthday

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Larimer, PhD, Principal Investigator — University of Washington
Locations (1):
- The Center for the Study of Health and Risk Behaviors, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No